CLINICAL TRIAL: NCT05259722
Title: A 24 Week, Randomised, Assessor Blinded, Active-controlled, Parallel Group, Phase 3, 2 Arm Trial to Compare the Efficacy and Safety of Delgocitinib Cream 20 mg/g Twice-daily With Alitretinoin Capsules Once-daily in Adult Participants With Severe Chronic Hand Eczema
Brief Title: A 24 Week Trial to Compare the Efficacy and Safety of Delgocitinib Cream 20 mg/g Twice-daily With Alitretinoin Capsules Once-daily in Adult Participants With Severe Chronic Hand Eczema
Acronym: DELTA FORCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0133-1528; 2021-003543-16 (EudraCT Number); U1111-1284-2242 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-02-18; First posted 2022-02-28 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hand Eczema
MeSH Terms: interventions — delgocitinib; Alitretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delgocitinib cream 20 mg/g (Experimental): Twice-daily topical application for up to 24 weeks
  Interventions: Drug: Delgocitinib
- Alitretinoin capsules 30 mg per capsule (Active Comparator): 1 capsule per day for up to 24 weeks
  Interventions: Drug: Toctino

INTERVENTIONS:
Drug: Delgocitinib — Cream for topical application 20 mg/g
  Arms: Delgocitinib cream 20 mg/g
Drug: Toctino — 1 capsule toctino 30 mg per day; optional reduction to 10 mg per day in case unacceptable adverse reactions to the higher dose occur
  Arms: Alitretinoin capsules 30 mg per capsule

SUMMARY:
This is a 24-week study in adult participants with severe chronic hand eczema (CHE) and with a documented inadequate response to treatment with topical corticosteroids (TCS) or for whom TCS are documented to be otherwise medically inadvisable. Eligible participants will be randomised to receive topical administration of delgocitinib cream 20 mg/g, twice-daily, or oral administration of alitretinoin capsules 30 mg (with an option to reduce to 10 mg during trial conduct), once-daily. The participants will visit the clinic regularly to have the study doctor assess their CHE and to answer questions about itch, pain, CHE symptoms, and quality of life.

The purpose of this trial is to compare the efficacy, health-related quality of life, and safety of delgocitinib cream and alitretinoin capsules.

ELIGIBILITY:
Main inclusion criteria:

* Diagnosis of CHE, defined as hand eczema that has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as severe at screening and baseline according to IGA-CHE (i.e. an IGA-CHE score of 4).
* Participants who have a documented recent history of inadequate response to treatment with topical corticosteroids (TCS) or for whom TCS are documented to be otherwise medically inadvisable (e.g. due to important side effects or safety risks).
* Participants adherent to standard non-medicated skin care including avoidance of known and relevant irritants and allergens.
* Participants must use contraceptive methods in accordance with local regulations regarding the methods of contraception for those participating in clinical studies

Main exclusion criteria:

* Concurrent skin diseases on the hands, e.g. tinea manuum.
* Active atopic dermatitis requiring medical treatment in regions other than the hands and feet.
* Active psoriasis on any part of the body.
* Hyperkeratotic hand eczema in combination with a history of psoriasis on any part of the body.
* Clinically significant infection on the hands.
* Participants who cannot receive alitretinoin.
* Clinically significant infection within 28 days prior to baseline which, in the opinion of the investigator, may compromise the safety of the participant in the trial, interfere with evaluation of the IMP, or reduce the participant's ability to participate in the trial.
* History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
* Any disorder which is not stable and could:

  * Affect the safety of the participant throughout the trial.
  * Impede the participant's ability to complete the trial.
* Positive hepatitis B surface antigen or hepatitis C virus antibody serology at screening.
* Systemic treatment with immunosuppressive drugs, immunomodulating drugs, retinoids, or corticosteroids within 28 days prior to baseline.
* Use of tanning beds, phototherapy, or bleach baths on the hands within 28 days prior to baseline.
* Previous or current treatment with Janus kinase (JAK) inhibitors (including delgocitinib/LEO 124249), systemic or topical.
* Cutaneously applied treatment with immunomodulators or TCS on the hands within 14 days prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 14 days prior to baseline.
* Other transdermal or cutaneously applied therapy on the hands (except for the use of subject's own emollients) within 7 days prior to baseline.
* Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 7 days prior to baseline.
* Treatment with any marketed biological therapy or investigational biologic agents:

  * Any cell-depleting agents: within 6 months prior to baseline, or until lymphocyte count returns to normal, whichever is longer.
  * Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to baseline.
* Previously used alitretinoin or participated in a clinical trial with alitretinoin or delgocitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (88):
- Austria (2):
  - LEO Pharma Investigational Site, Graz
  - LEO Pharma Investigational Site, Linz
- Canada (11):
  - LEO Pharma Investigational Site, Calgary
  - LEO Pharma Investigational Site, Edmonton
  - LEO Pharma Investigational Site, Guelph
  - LEO Pharma Investigational Site, London
  - LEO Pharma investigational site, London
  - LEO Pharma investigational site, Markham
  - LEO Pharma investigational site, Niagara Falls
  - LEO Pharma Investigational Site, North York
  - LEO Pharma investigational site, Québec
  - LEO Pharma Investigational Site, Red Deer
  - LEO Pharma investigational site, Sherbrooke
- France (7):
  - LEO Pharma Investigational Site, Antony
  - LEO Pharma Investigational Site, Martigues
  - LEO Pharma Investigational Site, Montpellier
  - LEO Pharma Investigational Site, Nice
  - LEO Pharma investigational site, Nice
  - LEO Pharma Investigational Site, Reims
  - LEO Pharma Investigational Site, Toulon
- Germany (24):
  - LEO Pharma Investigational Site, Augsburg
  - LEO Pharma Investigational Site, Berlin
  - LEO Pharma Investigational Site, Bochum
  - LEO Pharma Investigational Site, Bonn
  - LEO Pharma Investigational Site, Darmstadt
  - LEO Pharma Investigational Site, Dresden
  - LEO Pharma Investigational Site, Erlangen
  - LEO Pharma Investigational Site, Essen
  - LEO Pharma Investigational Site, Frankfurt
  - LEO Pharma Investigational Site, Friedrichshafen
  - LEO Pharma Investigational Site, Gera
  - LEO Pharma Investigational Site, Göttingen
  - LEO Pharma Investigational Site, Halle
  - LEO Pharma Investigational Site, Hamburg
  - LEO Pharma Investigational Site, Heidelberg
  - LEO Pharma Investigational Site, Langenau
  - LEO Pharma Investigational Site, Löhne
  - LEO Pharma Investigational Site, Mainz
  - LEO Pharma Investigational Site, Marburg
  - LEO Pharma Investigational Site, Memmingen
  - LEO Pharma Investigational Site, München
  - LEO Pharma Investigational Site, Oldenburg
  - LEO Pharma Investigational Site, Osnabrück
  - LEO Pharma Investigational Site, Wuppertal
- Italy (10):
  - LEO Pharma Investigational Site, Bologna
  - LEO Pharma Investigational Site, Brescia
  - LEO Pharma Investigational Site, Catania
  - LEO Pharma Investigational Site, Catanzaro
  - LEO Pharma Investigational Site, Genova
  - LEO Pharma Investigational Site, Lucca
  - LEO Pharma Investigational Site, Milan
  - LEO Pharma Investigational Site, Pavia
  - LEO Pharma Investigational Site, Pisa
  - LEO Pharma Investigational Site, Terracina
- Norway (2):
  - LEO Pharma Investigational Site, Stavanger
  - LEO Pharma Investigational Site, Tromsø
- Poland (15):
  - LEO Pharma Investigational Site, Bialystok
  - LEO Pharma investigational site, Bydgoszcz
  - LEO Pharma Investigational Site, Chorzów
  - LEO Pharma Investigational Site, Gdansk
  - LEO Pharma Investigational Site, Gdynia
  - LEO Pharma Investigational Site, Katowice
  - LEO Pharma investigational site, Katowice
  - LEO Pharma Investigational Site, Krakow
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Lublin
  - LEO Pharma Investigational Site, Poznan
  - LEO Pharma Investigational Site, Strzelce Opolskie
  - LEO Pharma Investigational Site, Szczecin
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw
- Slovakia (3):
  - LEO Pharma Investigational Site, Bratislava
  - LEO Pharma Investigational Site, Svidník
  - LEO Pharma Investigational Site, Trnava
- Spain (12):
  - LEO Pharma Investigational Site, Alcalá de Henares
  - LEO Pharma Investigational Site, Alicante
  - LEO Pharma Investigational Site, Badalona
  - LEO Pharma Investigational Site, Barcelona
  - LEO Pharma Investigational Site, Córdoba
  - LEO Pharma Investigational Site, L'Hospitalet de Llobregat
  - LEO Pharma Investigational Site, Madrid
  - LEO Pharma investigational site, Málaga
  - LEO Pharma investigational site, Pontevedra
  - LEO Pharma Investigational Site, Seville
  - LEO Pharma Investigational Site, Valencia
  - LEO Pharma Investigational Site, Zaragoza
- United Kingdom (2):
  - LEO Pharma Investigational Site, London
  - LEO Pharma Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gimenez-Arnau AM, Pinter A, Sondermann W, Reguiai Z, Woolf R, Lynde C, Legat FJ, Costanzo A, Silvestre JF, Mellerup N, Osterdal ML, Plohberger U, Ryttig L, Bauer A; trial investigators. Efficacy and safety of topical delgocitinib cream versus oral alitretinoin capsules in adults with severe chronic hand eczema (DELTA FORCE): a 24-week, randomised, head-to-head, phase 3 trial. Lancet. 2025 May 10;405(10490):1676-1688. doi: 10.1016/S0140-6736(25)00001-7. Epub 2025 Apr 16. PMID 40252681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled adult participants with severe CHE and with a documented inadequate response to treatment with TCS or for whom TCS were documented to be otherwise medically inadvisable.
Pre-assignment Details: Randomization was stratified by subtype (hyperkeratotic/non-hyperkeratotic) and region (North America/Europe).
Groups:
- Delgocitinib Cream 20 mg/g: Twice-daily topical application for up to 24 weeks.
  Delgocitinib: Cream for topical application 20 mg/g.
  There was a possibility to stop treatment after 16 weeks if IGA 0/1 was obtained.
- Alitretinoin Capsules 30 mg Per Capsule: 1 capsule per day for up to 24 weeks
  Toctino: 1 capsule toctino 30 mg per day; optional reduction to 10 mg per day in case unacceptable adverse reactions to the higher dose occur.
  There was a possibility to stop treatment after 12 weeks if IGA 0/1 was obtained.
Period: Overall Study
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Started | 254 | 259
Completed | 219 | 154
Not Completed | 35 | 105
Not completed — Adverse Event | 2 | 24
Not completed — Lost to Follow-up | 5 | 1
Not completed — Lack of Efficacy | 8 | 26
Not completed — Withdrawal by Subject | 15 | 33
Not completed — Various reasons | 3 | 9
Not completed — Not exposed to IMP | 1 | 12
Not completed — Discontinuation of IMP, related to COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Delgocitinib Cream 20 mg/g: Twice-daily topical application for up to 24 weeks>
  > Delgocitinib: Cream for topical application 20 mg/g
- Alitretinoin Capsules 30 mg Per Capsule: 1 capsule per day for up to 24 weeks>
  > Toctino: 1 capsule toctino 30 mg per day; optional reduction to 10 mg per day in case unacceptable adverse reactions to the higher dose occur
- Total: Total of all reporting groups
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule | Total
Number analyzed (Participants) | 254 | 259 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 238 | 233 | 471
  >=65 years | 16 | 26 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.78) | 44.0 (14.56) | 44.7 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 167 | 334
  Male | 87 | 92 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 14 | 36
  Not Hispanic or Latino | 226 | 241 | 467
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 237 | 240 | 477
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 29 | 54
  Austria | 2 | 3 | 5
  Norway | 1 | 1 | 2
  Poland | 89 | 91 | 180
  Italy | 13 | 9 | 22
  United Kingdom | 2 | 4 | 6
  Slovakia | 9 | 5 | 14
  France | 14 | 16 | 30
  Germany | 63 | 73 | 136
  Spain | 36 | 28 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in HECSI Score From Baseline to Week 12
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score) with a higher score indicating greater severity.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 249 | 250
score on a scale | -67.6 (3.37) | -51.5 (3.36)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; The change from baseline was analysed using an ANCOVA model with effects of treatment group, hyperkeratotic/non-hyperkeratotic subtype and baseline value of the score. Missing data was imputed with WOCF. Data after initiation of rescue treatment or permanent discontinuation of IMP was treated as missing; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -16.1, 95% CI 2-sided [-23.28 to -8.86]

2. Secondary Outcome: HECSI-90 at Week 12
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score), with a higher score indicating greater severity. HECSI-90 is defined as at least 90% improvement in HECSI score from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 249 | 250
Participants | 96 | 65
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; The difference in response rates was analysed using the Cochran-Mantel-Haenszel test stratified by hyperkeratotic/non-hyperkeratotic subtype. Missing data was imputed as non-response. Data after initiation of rescue treatment or permanent discontinuation of IMP was treated as missing; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.6, 95% CI 2-sided [4.34 to 20.78]

3. Secondary Outcome: IGA-CHE TS at Week 12.
Description: The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 250 | 253
Participants | 68 | 42
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.6, 95% CI 2-sided [3.31 to 17.87]

4. Secondary Outcome: Change in HESD Itch Score (Weekly Average) From Baseline to Week 12
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'itch' component.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 238 | 238
score on a scale | -3.0 (0.22) | -2.4 (0.21)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.12 to -0.20]

5. Secondary Outcome: Change in HESD Pain Score (Weekly Average) From Baseline to Week 12.
Description: The Hand Eczema Symptom Diary (HESD) is an eDiary in which participants will assess the worst severity of 6 individual signs and symptoms of CHE over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)' throughout the trial on a daily basis. This endpoint will only assess the 'pain' component.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 238 | 238
score on a scale | -2.9 (0.23) | -2.3 (0.23)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.018, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.08 to -0.10]

6. Secondary Outcome: AUC of HECSI-90 From Baseline up to Week 24
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score) with a higher score indicating greater severity. HECSI-90 is defined as at least 90% improvement in HECSI score from baseline. The area under the curve (AUC) at participant level will be determined as follows: 1 will be assigned when response is observed and 0 otherwise. The AUC is interpreted as number of days with 90% reduction in HECSI score until Week 24.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: days with 90% reduction in HECSI score
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 249 | 250
days with 90% reduction in HECSI score | 51.1 (4.11) | 43.5 (4.22)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; The AUC was analysed using a robust ANCOVA model with effects of treatment group, hyperkeratotic/non-hyperkeratotic subtype and baseline value of the score. Missing data was imputed as non-response. Data after initiation of rescue treatment or permanent discontinuation of IMP was treated as missing; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 14.3, 95% CI 2-sided [5.81 to 22.86]

7. Secondary Outcome: AUC of Change From Baseline in DLQI Score up to Week 24
Description: The Dermatology Life Quality Index (DLQI) is a validated questionnaire consisting of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their quality of life over the last week. The DLQI score is the sum of the 10 items (score ranging from 0 to 30); a high score is indicative of a poor quality of life. The area under the curve (AUC) at patient level will be determined from the change from baseline in DLQI score estimated as a piecewise linear function from Week 0 to Week 24. Differences will be analyzed with opposite sign to interpret positive area as improvement in scores and negative area as worsening.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: days * DLQI score reduction
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 230 | 236
days * DLQI score reduction | 1124.7 (61.37) | 790.7 (62.67)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; The AUC was analysed using a robust ANCOVA model with effects of treatment group, hyperkeratotic/non-hyperkeratotic subtype and baseline value of the score. Missing data was imputed with WOCF. Data after initiation of rescue treatment or permanent discontinuation of IMP was treated as missing; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 334.0, 95% CI 2-sided [195.69 to 472.26]

8. Secondary Outcome: Change in HECSI Score From Baseline to Week 24
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 249 | 250
score on a scale | -69.6 (3.78) | -45.1 (3.77)
Statistical Analysis 1: Comparison: Delgocitinib Cream 20 mg/g vs Alitretinoin Capsules 30 mg Per Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -24.5, 95% CI 2-sided [-32.55 to -16.36]

9. Secondary Outcome: Number of Treatment-emergent AEs From Baseline up to Week 26
Description: An adverse event (AE) will be considered treatment emergent if started after the first application of investigational medicinal product (IMP), or if started before the first application of IMP and worsened in severity after first dose of IMP.
Time Frame: 26 weeks
Measure: Number; unit: events
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 253 | 247
events | 280 | 620

10. Secondary Outcome: Number of Treatment-emergent SAEs From Baseline up to Week 26
Description: A serious adverse event (SAE) will be considered treatment emergent if started after the first application of investigational medicinal product (IMP), or if started before the first application of IMP and worsened in severity after first dose of IMP.
Time Frame: 26 weeks
Measure: Number; unit: events
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 253 | 247
events | 5 | 12

11. Secondary Outcome: Number of AEs Leading to IMP Discontinuation up to Week 24
Description: The investigational medicinal product (IMP) will be discontinued permanently in case of an AE that, in the opinion of the investigator or sponsor's medical expert, contraindicates further dosing. The investigator will assess the relationship between investigational medicinal product (IMP) and the adverse event (AE).
Time Frame: 24 weeks
Measure: Number; unit: events
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
Number analyzed (Participants) | 253 | 247
events | 4 | 44

ADVERSE EVENTS:
Time Frame: From baseline to Week 26
Groups:
- Delgocitinib Cream 20 mg/g: Delgocitinib Cream 20 mg/g (N=253)
- Alitretinoin Capsules 30 mg Per Capsule: Alitretinoin Capsules 30 mg Per Capsule (N=247)
Arm/Group | Delgocitinib Cream 20 mg/g | Alitretinoin Capsules 30 mg Per Capsule
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/247
Serious Adverse Events (participants affected / at risk) | 5/253 | 12/247
Other Adverse Events (participants affected / at risk) | 58/253 | 143/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 20 mg/g (N=253) | Alitretinoin Capsules 30 mg Per Capsule (N=247)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 20 mg/g (N=253) | Alitretinoin Capsules 30 mg Per Capsule (N=247)
Dry eye (Eye disorders) | 0 (0) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Lip dry (Gastrointestinal disorders) | 0 (0) | 8 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 14 (15)
COVID-19 (Infections and infestations) | 5 (5) | 9 (9)
Nasopharyngitis (Infections and infestations) | 30 (38) | 34 (46)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 8 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 10 (11)
Blood triglycerides increased (Investigations) | 2 (2) | 7 (8)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 10 (19) | 79 (113)
Migraine (Nervous system disorders) | 2 (2) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (10)
Flushing (Vascular disorders) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT05259722/Prot_SAP_000.pdf